CLINICAL TRIAL: NCT01573988
Title: Behavioural and Metabolic Consequences of Increasing Eating Frequency
Brief Title: Satiety, Meal Frequency and Nutritional Aspects
Acronym: SAFRAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting of volunteers with a BMI (Body Mass Index) between 30 and 35 kg/m2
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010.612/16
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Volunteers
Keywords: Nutrition; Eating frequency; Food intake; Eating behavior; Satiety; Ghrelin
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-obese volunteers (Other): Volunteers with a BMI (Body Mass Index) between 20 and 25 kg/m2.
  Interventions: Other: Increasing eating frequency
- Obese volunteers (Other): Volunteers with a BMI (Body Mass Index) between 30 and 35 kg/m2.
  Interventions: Other: Increasing eating frequency

INTERVENTIONS:
Other: Increasing eating frequency — The subjects receive the same breakfast with two sequences :
  * breakfast in one intake at 8:00
  * breakfast in four isocaloric intakes (8:00, 9:00, 10:00, 11:00) The sequence made twice : one for metabolic study and one for the study of eating behavior
  The lunch during metabolic study is a standard meal The lunch during behavioural study is an ad libitum buffet test meal.
  The administration order is determined by randomized allocation. The wash-out period is one to three weeks.
  There are not diet or exercise interventions.

SUMMARY:
In this study, the investigators are interested in assessing the effects of the isocaloric increase of eating frequency on appetite and metabolism. How the consumption of an isocaloric breakfast in four intakes vs. one can modify satiety and appetite control in lean and obese subjects through :

* the physiological consequences : difference in postprandial kinetics of glucose, non esterified fatty acid, triglyceride, the secretion of satiety gut hormone (insulin, ghrelin, leptin and cholescystokinine (CCK), peptide YY (PYY), glucagon-like peptide-1 (GLP-1), nutrients oxidative fate and plasmatic oxidative stress (Malondialdehyde (MDA), glutathion, lipid hydroperoxides)
* eating behavior during an ad libitum buffet test meal

ELIGIBILITY:
Inclusion Criteria:

* No smokers
* BMI 20 to 35 kg/m2
* Moderate physical activity
* Safety during medical consultation
* Feeding behavioural phenotype (Dutch Eating Questionnaire, Three Eating Factor Questionnaire)

Exclusion Criteria:

* Medical history which may affect glucose metabolism (diabetes, renal or hepatic failure, thyroid dysfunction, Cushing syndrome, acromegaly…)
* Medical history which affect nutrient absorption (gastro-intestinal and pancreatic disease, gastrectomy, colectomy…)
* Drug use in the last two months that could affect glucose metabolism (steroids, topical gastric preparation, anorectic drugs…)
* Eating disorders
* Claustrophobic subjects

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ghrelin plasmatic concentration | 240 minutes after breakfast beginning (just before the lunch)

SECONDARY OUTCOMES:
Satiety through food intakes (quantitative) at the ad libitum buffet test meal | Since the beginning of the buffet test meal (240 minutes after breakfast beginning) to the end of the meal (at the latest 270 minutes after breakfast beginning).
Satiety through visual analogue scale | 240 minutes after breakfast beginning (just before the lunch)
Plasma metabolite concentrations (glycaemia, non esterified fatty acid, | kinetics during 430 minutes
Endocrine concentrations (insulin, ghrelin, GLP-1, PYY, leptin, C-peptide) | kinetics during 430 minutes
Plasma markers of oxidative stress (MDA, gluthation, lipid hydroxide) | kinetics during 430 minutes
Lipid oxidation | kinetics during 430 minutes
Eating behaviour at the buffet test meal by video recording (food choice, nutritional composition of the meal , kinetics of nutrient intake, meal structure, lunch duration) | during the buffet test meal (max : 30 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud - Centre de Recherche en Nutrition Humaine, Pierre-Bénite, France

REFERENCES:
- See also: Related Info — http://www.crnh-rhone-alpes.fr/spip.php?article145&idprojet=22